CLINICAL TRIAL: NCT04210986
Title: Senolytic Drugs Attenuate Osteoarthritis-Related Articular Cartilage Degeneration: A Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Steadman Philippon Research Institute (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-16
Record Dates: First submitted 2019-12-03; First posted 2019-12-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
Keywords: Fisetin; Inflammation; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation; Osteoarthritis | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fisetin (Experimental): Fisetin 100 mg capsules (~20 mg/ kg/ day) will be administered orally for two consecutive days (days 1 and 2) followed by 28 days off. A second course will be given for two consecutive days (days 31 and 32)
  Interventions: Dietary Supplement: Fisetin
- Placebo (Placebo Comparator): Placebo capsules will be administered orally for two consecutive days (days 1 and 2) followed by 28 days off. A second course will be given for two consecutive days (days 31 and 32)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: Fisetin — Fisetin will be administered orally at 20 mg/kg for two consecutive days, followed by 28 days off, then 2 more consecutive days.
  Other Names: Novusetin; 7,3',4'-flavon-3-ol; 3,3',4',7-tetrahydroxyflavone
  Arms: Fisetin
Drug: Placebo oral capsule — Placebo will be administered orally for two consecutive days, followed by 28 days off, then 2 more consecutive days.
  Other Names: Inactive drug
  Arms: Placebo

SUMMARY:
Phase I/II randomized, double-blind, placebo-controlled clinical trial to test the safety and efficacy of Fisetin for treating mild to moderate osteoarthritis

DETAILED DESCRIPTION:
This is a Phase I/II randomized, double-blind, placebo-controlled clinical trial that will be conducted at The Steadman Clinic (TSC) and Steadman Philippon Research Institute (SPRI). The purpose of this study is to evaluate the clinical efficacy of Fisetin (FIS), a dietary supplement, in symptomatic knee osteoarthritis (OA) patients. Key aspects of this proposal include the investigator's well-developed methodologies to measure and compare systemic senescence-associated secretory phenotype (SASP) including inflammatory biomarkers and senescent cells, and collect magnetic resonance images, self-reported outcomes, physical performance and other objective clinical data. Given the drug FIS has been empirically demonstrated to reduce senescent cell burden, the main objective(s) are to determine 1) the safety of FIS during dosing and 2) whether FIS reduces senescent cells, pro-inflammatory and cartilage degenerating SASP markers, and reduces OA-symptoms leading to improved joint health and function.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be included if all the following criteria are met:

1. Are male or female, ages 40-80;
2. Are willing to comply with all study related procedures and assessments;
3. Are ambulatory as defined by ability to complete functional performance testing;
4. Radiographic evidence of Kellgren-Lawrence grade II-IV osteoarthritis in one or both knees;
5. Scores 4-10 on the Numerical Rating Scale (NRS) for pain;
6. Stable dose of screening/baseline medications for at least 2 months prior to the anticipated date of study drug dosing.

Exclusion Criteria:

Subjects will be excluded if any of the following criteria are met:

1. Females who are nursing, pregnant or planning to become pregnant during the duration of study drug dosing;
2. Males who do not wish to abstain from sex or use contraceptive protection during study drug dosing and for 2 weeks after the last dose;
3. Subjects who do not have the capacity to consent themselves;
4. Subjects who are unable to tolerate oral medication;
5. Subjects having previously undergone any of the following treatments in the stated time window.

   * Surgery on the Study Knee in the past 6 months;
   * Partial or complete joint replacement in the study knee. Partial or complete joint replacement in the contralateral knee is acceptable as long as the surgery was performed at least 6 months prior to enrollment and the operative knee is asymptomatic;
   * Patients who have undergone arthroscopic surgery (including microfracture and meniscectomy) on the Study Knee in the last 2 years prior to the Screening visit or are anticipated to have arthroscopic surgery on either knee at any time during the study period;
   * Steroid injection, including extended-release corticosteroid (e.g., Zilretta®) within the last 5 months;
   * Biologic (platelet-rich plasma, bone marrow, adipose tissue/cells) or hyaluronic acid injection into the Study Knee in the past 6 months;
6. Subjects with any of the following drug/medication statuses:

   * Currently taking Losartan;
   * Currently taking Warfarin or related anticoagulants;
   * Opioid analgesics taken in the past 8 weeks and are not willing to discontinue these medications through the duration of the study;
   * Senolytic agents taken within the past 6 months and are not willing to discontinue these medications through the duration of the study, including: Fisetin, Quercetin, Luteolin, Dasatinib, Piperlongumine, or Navitoclax;
   * Drugs that induce significant cellular stress and are not willing to discontinue these medications through the duration of the study, including alkylating agents, anthracyclines, platins, other chemotherapy drugs;
   * Subjects taking the following other drugs if they cannot be held (per the Principal Investigator) for at least 2 days before and during administration of Fisetin: cyclosporine, tacrolimus, repaglinide, and bosentan.
7. Subjects with any of the following disease statuses:

   * Significant liver disease (i.e. greater than or equal to 2x the upper limit of normal bilirubin levels) or as in the opinion of the Principal Investigator;
   * Significant renal disease (eGFR of <60 ml/min/1.73m2) or as in the opinion of the Principal Investigator;
   * History of other formally diagnosed joint diseases including osteonecrosis, acromegaly, Paget's disease, Ehlers-Danlos Syndrome, Gaucher's disease, Cushing's syndrome, Stickler's syndrome, joint infection, hemophilia, hemochromatosis, or neuropathic arthropathy of any cause;
   * Any active systemic autoimmune disease with musculoskeletal involvement or any history of system inflammatory arthritis;
   * Patients with type 1 or 2 diabetes (HbA1c>6.5%) and/or taking medications that affect insulin levels, including: Metformin (within the last week), Glucocorticoids (within the last month), Acarbose (within the last week);
8. Subjects unable to safely practically undergo an MRI (BMI > 40 kg/m2) or size exceeding limits of MRI equipment, implanted metal in study knee near joint surface, incompatible implant/device, severe claustrophobia;
9. Subjects that have any medical condition, including laboratory findings and findings in the medical history or in the pre-study assessments, that in the opinion of the Investigator constitutes a risk or contraindication for participation in the study or that could interfere with the study objectives, conduct or evaluation or prevent the patient from fully participating in all aspects of the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Evans, MD, Principal Investigator — The Steadman Clinic
Locations (1):
- The Steadman Clinic, Vail, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fisetin | Placebo
Started | 34 | 40
Completed (Protocol completion defined as completion of the final in-person and/or remote assessment, or knowledge of conversion to an alternative treatment modality as defined in the protocol.) | 25 | 35
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fisetin | Placebo | Total
Number analyzed (Participants) | 34 | 40 | 74
Age, Continuous [Median (Full Range); unit: years] | 62 [44 to 77] | 64 [42 to 79] | 63 [42 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 14 | 16 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 33 | 39 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 34 | 38 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 34 | 40 | 74

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing One or More Treatment-Emergent Adverse Event
Description: Number of Participants Experiencing one or more Treatment-Emergent Adverse Event (TEAE) within each group.
Time Frame: Duration of study, an average of 12 months
Population: All participants randomized and dosed with study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
Participants | 28 | 33
Statistical Analysis 1: Comparison: Fisetin vs Placebo; Null hypothesis: no difference in proportion of participants experiencing any TEAE between Fisetin and Placebo groups; Test type: Superiority; p > 0.9, Fisher Exact — No adjustment made for multiple comparisons; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.25 to 4.02] — Odds ratio is for fisetin group, relative to the placebo group

2. Secondary Outcome: Change in Levels of Pro-inflammatory Markers Associated With Senescence
Description: Serum C-reactive protein (CRP) level measured on ELISA. The enzyme linked immunoassay (ELISA) is a laboratory technique that detects certain antigens in the blood. ELISA was used to detect the level of CRP in the blood. The liver releases CRP into blood in response to inflammation. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 14 days, 45 days, 6 months, 12 months (post 1st drug dose)
Population: The analysis dataset is comprised of all randomized study participants with an evaluable endpoint data captured at each assessment time point. Unavailability of endpoint data at post-intervention time points may be due to withdrawal, discontinuation, missed study visit, or otherwise unsuccessful data acquisition or processing.
Measure: Least Squares Mean (Standard Error); unit: ug/ml
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
ug/ml
  C-reactive protein (CRP): Day 14: number analyzed (Participants) | 29 | 30
  C-reactive protein (CRP): Day 14 | 14.0 (2.5) | 10.5 (2.5)
  C-reactive protein (CRP): Day 45: number analyzed (Participants) | 29 | 34
  C-reactive protein (CRP): Day 45 | 8.9 (1.9) | 6.4 (1.8)
  C-reactive protein (CRP): Month 6: number analyzed (Participants) | 27 | 33
  C-reactive protein (CRP): Month 6 | 32.5 (6.4) | 12.0 (5.7)
  C-reactive protein (CRP): Month 12: number analyzed (Participants) | 24 | 31
  C-reactive protein (CRP): Month 12 | 9.2 (1.8) | 8.8 (1.6)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; DAY 14 ASSESSMENT Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p = 0.9728, Mixed Models Analysis — A priori threshold for statistical significance = 0.05. P-values adjusted for the number of post-intervention assessments via Holm-Bonferroni method; Mixed model for repeated measures (mmrm). Baseline measurement included as covariate. Random intercept and slope. Kenward-Roger DF; Contrast of LS Means = -3.5, 95% CI 2-sided [-10.6 to 3.6] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; DAY 45 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p = 0.9728, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -2.5, 95% CI 2-sided [-7.8 to 2.8] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 3: Comparison: Fisetin vs Placebo; MONTH 6 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p = 0.0829, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -20.5, 95% CI 2-sided [-37.7 to -3.3] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 4: Comparison: Fisetin vs Placebo; MONTH 12 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p = 0.9728, Contrast of LS Means — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.5 — Direction of Estimation Parameter: Placebo - Fisetin

3. Secondary Outcome: Change in Levels of Cartilage Degenerating Markers Associated With OA
Description: Serum cartilage oligomeric matrix protein (COMP) level measured on ELISA. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 14 days, 45 days, 6 months, 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
ng/ml
  COMP: Day 14: number analyzed (Participants) | 34 | 38
  COMP: Day 14 | 288.3 (19.0) | 290.1 (17.5)
  COMP: Day 45: number analyzed (Participants) | 31 | 39
  COMP: Day 45 | 274.2 (18.1) | 285.2 (15.6)
  COMP: Month 6: number analyzed (Participants) | 26 | 34
  COMP: Month 6 | 282.0 (22.0) | 241.7 (18.2)
  COMP: Month 12: number analyzed (Participants) | 22 | 26
  COMP: Month 12 | 274.9 (14.1) | 268.0 (12.7)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; DAY 14 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 2.52, 95% CI 2-sided [-49.4 to 54.5] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 11.0, 95% CI 2-sided [-36.8 to 58.8] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 3: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.6594, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -40.3, 95% CI 2-sided [-97.6 to 17.1] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 4: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -6.9, 95% CI 2-sided [-45.5 to 31.7] — Direction of Estimation Parameter: Placebo - Fisetin

4. Secondary Outcome: Change in Physical Function of the Study Knee (6 Min Walk)
Description: The 6 minute walk test (6MWT) assesses distance (in meters) walked over 6 minutes as a sub-maximal test of aerobic capacity, exercise tolerance and endurance. The score range for healthy adults is 400-700 m, depending on age and sex. Shorter distances indicate increased impairment. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
Meters
  Walk Distance: Month 6: number analyzed (Participants) | 29 | 36
  Walk Distance: Month 6 | 541.8 (8.7) | 552.2 (7.8)
  Walk Distance: Month 12: number analyzed (Participants) | 25 | 31
  Walk Distance: Month 12 | 544.2 (8.0) | 543.6 (7.2)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.7480, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 10.5, 95% CI 2-sided [-12.9 to 33.9] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.9572, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.6, 95% CI 2-sided [-22.2 to 21.1] — Direction of Estimation Parameter: Placebo - Fisetin

5. Secondary Outcome: Change in Physical Function of the Study Knee (Timed-up-and-go Test)
Description: The Timed Up and Go (TUG) test measures how long it takes (in seconds) to stand up, walk a distance of 10 feet, turn, walk back, and sit down again. < 10 seconds is considered normal. Longer times indicate poorer function. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
seconds
  Up and go time: Month 6: number analyzed (Participants) | 29 | 36
  Up and go time: Month 6 | 6.08 (0.18) | 6.09 (0.16)
  Up and go time: Month 12: number analyzed (Participants) | 25 | 31
  Up and go time: Month 12 | 5.93 (0.15) | 6.00 (0.13)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.01, 95% CI 2-sided [-0.47 to 0.49] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.07, 95% CI 2-sided [-0.33 to 0.47] — Direction of Estimation Parameter: Placebo - Fisetin

6. Secondary Outcome: Change in Physical Function of the Study Knee (Fast 4-meter Walk)
Description: fast 4-meter walk test (4MW). The 4MW was assessed at the fastest safe speed for each participant. This test assesses the capacity for performance of certain activities (e.g., crossing a street before the light changes). Units are m/s, and slower speeds indicate greater impairment. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: meters/second
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
meters/second
  Walk Time: Month 6: number analyzed (Participants) | 29 | 36
  Walk Time: Month 6 | 22.1 (0.46) | 21.7 (0.41)
  Walk Time: Month 12: number analyzed (Participants) | 25 | 31
  Walk Time: Month 12 | 21.7 (0.36) | 21.8 (0.32)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.37, 95% CI 2-sided [-1.61 to 0.87] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.16, 95% CI 2-sided [-0.80 to 1.13] — Direction of Estimation Parameter: Placebo - Fisetin

7. Secondary Outcome: Change in Physical Function of the Study Knee (LEK)
Description: Peak knee adduction moment (KAM) during stance phase of gait in the affected leg, determined using video-motion analysis and force plate data. Values are normalized by mass*height of participant. Higher KAM has been associated with more rapid osteoarthritis progression. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Newton*meter / (kilogram*meter)
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
Newton*meter / (kilogram*meter)
  Adduction Moment (affected): Month 6: number analyzed (Participants) | 29 | 36
  Adduction Moment (affected): Month 6 | 0.204 (0.009) | 0.182 (0.008)
  Adduction Moment (affected): Month 12: number analyzed (Participants) | 24 | 30
  Adduction Moment (affected): Month 12 | 0.204 (0.009) | 0.180 (0.009)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.130, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.022, 95% CI 2-sided [-0.045 to 0.002] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.130, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.024, 95% CI 2-sided [-0.049 to 0.002] — Direction of Estimation Parameter: Placebo - Fisetin

8. Secondary Outcome: Change in Physical Function of the Study Knee (Stair-Climbing Test)
Description: The Stair-Climbing Test assesses the time required (in seconds) to ascend and descend a standard flight of 10 stairs. Longer times indicate poorer physical function. Stairs require greater knee extensor force than gait, so this test may be more sensitive to osteoarthritis pain and function than walking tests. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
seconds
  Stairs Time: Month 6: number analyzed (Participants) | 29 | 36
  Stairs Time: Month 6 | 8.88 (0.23) | 8.66 (0.21)
  Stairs Time: Month 12: number analyzed (Participants) | 25 | 31
  Stairs Time: Month 12 | 8.66 (0.30) | 8.78 (0.27)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.9584, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.22, 95% CI 2-sided [-0.84 to 0.40] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.9584, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.12, 95% CI 2-sided [-0.69 to 0.92] — Direction of Estimation Parameter: Placebo - Fisetin

9. Secondary Outcome: Change in Muscle Strength (Isokinetic Dynamometry)
Description: This test utilizes an isokinetic dynamometer to assess the peak knee extension torque that can be produced by the affected leg at a constant rate of knee extension (60 degrees/s). The resulting measure is normalized by body mass and reported with units Newton-meters (Nm). Increased torque over time would indicate improved muscle strength and/or decreased joint pain. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Newton-meters (Nm)
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
Newton-meters (Nm)
  Quad Torque (affected): Month 6: number analyzed (Participants) | 29 | 36
  Quad Torque (affected): Month 6 | 81.2 (2.6) | 83.1 (2.3)
  Quad Torque (affected): Month 12: number analyzed (Participants) | 24 | 29
  Quad Torque (affected): Month 12 | 81.2 (2.6) | 85.0 (2.3)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.5905, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 1.88, 95% CI 2-sided [-5.07 to 8.84] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.5414, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 3.86, 95% CI 2-sided [-3.08 to 10.79] — Direction of Estimation Parameter: Placebo - Fisetin

10. Secondary Outcome: Evaluation of Patient Reported Outcomes (PROs) for Knee Pain
Description: Numeric Rating Scale (NRS) reporting 'pain today'. Scale of 0-10 with 0 representing 'no pain' and 10 representing 'severe pain'. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: every 3 days for the first 6-weeks of drug dosing, then weekly for an additional 6 weeks.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
score on a scale
  NRS Pain Today: Day 3: number analyzed (Participants) | 25 | 30
  NRS Pain Today: Day 3 | 2.80 (0.29) | 2.85 (0.27)
  NRS Pain Today: Day 6: number analyzed (Participants) | 28 | 32
  NRS Pain Today: Day 6 | 2.43 (0.33) | 2.87 (0.30)
  NRS Pain Today: Day 9: number analyzed (Participants) | 23 | 30
  NRS Pain Today: Day 9 | 2.35 (0.41) | 2.77 (0.37)
  NRS Pain Today: Day 12: number analyzed (Participants) | 27 | 32
  NRS Pain Today: Day 12 | 2.47 (0.31) | 2.40 (0.28)
  NRS Pain Today: Day 15: number analyzed (Participants) | 30 | 32
  NRS Pain Today: Day 15 | 2.65 (0.37) | 2.18 (0.35)
  NRS Pain Today: Day 18: number analyzed (Participants) | 23 | 30
  NRS Pain Today: Day 18 | 2.58 (0.36) | 2.39 (0.32)
  NRS Pain Today: Day 21: number analyzed (Participants) | 26 | 36
  NRS Pain Today: Day 21 | 2.25 (0.29) | 2.44 (0.26)
  NRS Pain Today: Day 24: number analyzed (Participants) | 29 | 32
  NRS Pain Today: Day 24 | 2.46 (0.32) | 2.57 (0.29)
  NRS Pain Today: Day 27: number analyzed (Participants) | 28 | 34
  NRS Pain Today: Day 27 | 2.35 (0.28) | 2.36 (0.25)
  NRS Pain Today: Day 30: number analyzed (Participants) | 29 | 37
  NRS Pain Today: Day 30 | 2.58 (0.30) | 2.21 (0.27)
  NRS Pain Today: Day 33: number analyzed (Participants) | 30 | 27
  NRS Pain Today: Day 33 | 2.09 (0.29) | 2.19 (0.27)
  NRS Pain Today: Day 36: number analyzed (Participants) | 25 | 35
  NRS Pain Today: Day 36 | 2.57 (0.30) | 2.37 (0.27)
  NRS Pain Today: Day 39: number analyzed (Participants) | 27 | 29
  NRS Pain Today: Day 39 | 2.15 (0.30) | 2.26 (0.27)
  NRS Pain Today: Day 42: number analyzed (Participants) | 22 | 35
  NRS Pain Today: Day 42 | 2.42 (0.28) | 1.81 (0.24)
  NRS Pain Today: Week 7: number analyzed (Participants) | 29 | 36
  NRS Pain Today: Week 7 | 2.15 (0.29) | 1.92 (0.26)
  NRS Pain Today: Week 8: number analyzed (Participants) | 28 | 35
  NRS Pain Today: Week 8 | 2.04 (0.25) | 1.84 (0.23)
  NRS Pain Today: Week 9: number analyzed (Participants) | 30 | 33
  NRS Pain Today: Week 9 | 1.84 (0.24) | 1.86 (0.22)
  NRS Pain Today: Week 10: number analyzed (Participants) | 26 | 31
  NRS Pain Today: Week 10 | 1.88 (0.29) | 1.71 (0.26)
  NRS Pain Today: Week 11: number analyzed (Participants) | 28 | 34
  NRS Pain Today: Week 11 | 1.99 (0.28) | 1.57 (0.25)
  NRS Pain Today: Week 12: number analyzed (Participants) | 30 | 32
  NRS Pain Today: Week 12 | 2.26 (0.39) | 1.91 (0.36)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; DAY 3 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.05, 95% CI 2-sided [-0.75 to 0.85] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; DAY 6 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.44, 95% CI 2-sided [-0.45 to 1.34] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 3: Comparison: Fisetin vs Placebo; DAY 9 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.42, 95% CI 2-sided [-0.70 to 1.54] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 4: Comparison: Fisetin vs Placebo; DAY 12 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.06, 95% CI 2-sided [-0.91 to 0.78] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 5: Comparison: Fisetin vs Placebo; DAY 15 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.47, 95% CI 2-sided [-1.50 to 0.56] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 6: Comparison: Fisetin vs Placebo; DAY 18 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.19, 95% CI 2-sided [-1.16 to 0.77] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 7: Comparison: Fisetin vs Placebo; DAY 21 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.19, 95% CI 2-sided [-0.58 to 0.96] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 8: Comparison: Fisetin vs Placebo; DAY 24 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.10, 95% CI 2-sided [-0.76 to 0.97] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 9: Comparison: Fisetin vs Placebo; DAY 27 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.01, 95% CI 2-sided [-0.74 to 0.76] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 10: Comparison: Fisetin vs Placebo; DAY 30 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.38, 95% CI 2-sided [-1.20 to 0.44] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 11: Comparison: Fisetin vs Placebo; DAY 33 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.10, 95% CI 2-sided [-0.69 to 0.89] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 12: Comparison: Fisetin vs Placebo; DAY 36 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.20, 95% CI 2-sided [-1.02 to 0.61] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 13: Comparison: Fisetin vs Placebo; DAY 39 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.11, 95% CI 2-sided [-0.70 to 0.92] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 14: Comparison: Fisetin vs Placebo; DAY 42 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.62, 95% CI 2-sided [-1.36 to 0.13] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 15: Comparison: Fisetin vs Placebo; WEEK 7 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.23, 95% CI 2-sided [-1.01 to 0.55] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 16: Comparison: Fisetin vs Placebo; WEEK 8 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.20, 95% CI 2-sided [-0.89 to 0.49] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 17: Comparison: Fisetin vs Placebo; WEEK 9 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.02, 95% CI 2-sided [-0.63 to 0.67] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 18: Comparison: Fisetin vs Placebo; WEEK 10 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.17, 95% CI 2-sided [-0.95 to 0.61] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 19: Comparison: Fisetin vs Placebo; WEEK 11 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.42, 95% CI 2-sided [-1.18 to 0.34] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 20: Comparison: Fisetin vs Placebo; WEEK 12 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.35, 95% CI 2-sided [-1.41 to 0.71] — Direction of Estimation Parameter: Placebo - Fisetin

11. Secondary Outcome: Evaluation of Patient Reported Outcomes (PROs) for Knee Function
Description: Western Ontario and McMaster Universities Arthritis Index (WOMAC) - total score. Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status. The higher the score, the poorer the function. All post-intervention group comparisons were adjusted for the baseline value as a covariate.
Time Frame: 6 months, 12 months, and 18 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
score on a scale
  WOMAC Total: Month 6: number analyzed (Participants) | 28 | 34
  WOMAC Total: Month 6 | 15.2 (1.8) | 17.1 (1.7)
  WOMAC Total: Month 12: number analyzed (Participants) | 21 | 26
  WOMAC Total: Month 12 | 19.6 (2.1) | 15.4 (1.9)
  WOMAC Total: Month 18: number analyzed (Participants) | 19 | 23
  WOMAC Total: Month 18 | 17.4 (2.0) | 17.4 (1.8)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 3]; Test type: Superiority; p = 0.9106, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 1.86, 95% CI 2-sided [-3.09 to 6.82] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; [analysis description as in outcome 2, analysis 4]; Test type: Superiority; p = 0.4424, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -4.20, 95% CI 2-sided [-9.93 to 1.53] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 3: Comparison: Fisetin vs Placebo; MONTH 18 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment; Test type: Superiority; p = 0.9901, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -0.03, 95% CI 2-sided [-5.55 to 5.48] — Direction of Estimation Parameter: Placebo - Fisetin

12. Secondary Outcome: Change in the Quality of Articular Cartilage in the Study Knee With Quantitative Magnetic Resonance Imaging (MRI)
Description: Mean T2 relaxation times were determined across 4 subregions: central medial femur (CMF), central lateral femur (CLF), central medial tibia (CMT), and central lateral tibia (CLT). All post-intervention group comparisons were adjusted for the baseline value as a covariate. The mean T2 changes over time for all subregions were listed in rank order from most positive (indicating worsened cartilage condition over time) to most negative (indicating improved cartilage condition over time). These unitless rankings were used in a Sum of Ranks statistical analysis to compare cartilage changes across different knee joint regions without assuming normality (as appropriate for MRI data). There are no published standards for what would be considered a clinically significant effect for sum-of-ranks cartilage T2 data, so it was assumed that a statistically significant difference would imply clinical significance as well.
Time Frame: 6 months, and 12 months (post 1st drug dose)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Unitless
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
Unitless
  Sum of Ranks Mean T2: Month 6: number analyzed (Participants) | 28 | 34
  Sum of Ranks Mean T2: Month 6 | 149.6 (11.6) | 150.3 (10.7)
  Sum of Ranks Mean T2: Month 12: number analyzed (Participants) | 24 | 30
  Sum of Ranks Mean T2: Month 12 | 156.1 (13.0) | 144.8 (12.0)
Statistical Analysis 1: Comparison: Fisetin vs Placebo; MONTH 6 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment. A priori power calculation was based a standardized mean difference effect size of SMD=0.73 (Mackay, et al, 2018, Osteoarthritis and Cartilage); Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = 0.69, 95% CI 2-sided [-30.95 to 32.3] — Direction of Estimation Parameter: Placebo - Fisetin
Statistical Analysis 2: Comparison: Fisetin vs Placebo; MONTH 12 ASSESSMENT. Null hypothesis: no difference in baseline-adjusted least squares means between Fisetin and Placebo groups at each post-intervention assessment. A priori power calculation was based a standardized mean difference effect size of SMD=0.73 (Mackay, et al, 2018, Osteoarthritis and Cartilage); Test type: Superiority; p > 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Contrast of LS Means = -11.3, 95% CI 2-sided [-46.9 to 24.2] — Direction of Estimation Parameter: Placebo - Fisetin

13. Secondary Outcome: Number of Participants Who Convert to Alterative Treatment Within Each Group.
Description: Patients will be allowed to receive a steroid injection and still participate in the study. All participants that undergo alternative therapy (e.g. total knee arthroplasty or biologic injection) will be recorded, and proportions will be compared between groups.
Time Frame: Any time during 18-month monitoring period.
Population: The analysis dataset is comprised of all randomized study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Fisetin | Placebo
Number analyzed (Participants) | 34 | 40
Participants | 1 | 3
Statistical Analysis 1: Comparison: Fisetin vs Placebo; With only 4 participants that converted to an alternative treatment modality, this analysis is underpowered; Test type: Superiority; p = 0.474, Log Rank — A priori threshold for statistical significance = 0.05; Cox proportional hazards model constructed. Score (log rank) test to assess between group difference in hazard rate; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.05 to 4.21] — Hazard ratio expresses the hazard rate of the Fisetin group in the numerator and the hazard rate of the Placebo group in the denominator

ADVERSE EVENTS:
Time Frame: 12 months following initial administration of study medication.
Description: AE assessment occurred systematically at in-person visits at 14 days, 45 days, 6 months, and 12 months following first dose.
  Additionally, dosing reminder phone calls occurred at the time of subsequent dosing, at which time AEs were captured.
Arm/Group | Fisetin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/40
Serious Adverse Events (participants affected / at risk) | 2/34 | 2/40
Other Adverse Events (participants affected / at risk) | 28/34 | 33/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fisetin (N=34) | Placebo (N=40)
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Rotator cuff repair secondary to massive rotator cuff tear.
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Low back pain treated with lumbar microdiscectomy.
Bladder Perforation (Renal and urinary disorders) | 1 (1) | 0 (0) — Iatrogenic bladder injury during hip replacement surgery.
Tracheal Stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Surgery for subglottic stenosis.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fisetin (N=34) | Placebo (N=40)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (17) | 17 (23)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (5)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Dry Mouth (Gastrointestinal disorders) | 2 (3) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Lab Findings (General disorders) | 4 (8) | 3 (5)
Fatigue (General disorders) | 3 (3) | 3 (3)
Covid 19 (General disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 2 (3)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (5)
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04210986/Prot_SAP_ICF_002.pdf